CLINICAL TRIAL: NCT07032116
Title: Evidence-based Evaluation of Yiqi Jiangzhuo Huoxue Tongluo Method in Delaying the Occurrence of End-stage Renal Disease in Diabetic Kidney Disease--Study 1
Brief Title: YiqiJiangzhuoHuoxueTongluo Method to Delay the Occurrence of End-stage Renal Disease in Diabetic Kidney Disease--Study1
Status: Not yet recruiting | Type: Observational
Sponsor: Liu Hongfang (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Tianjin Medical University Chu Hsien-I Memorial Hospital (Unknown); Changchun University of Chinese Medicine (Other); EFONG PHARMRCEUTICRL (Unknown); Xinxiang Central Hospital of Henan province (Unknown); Xiamen Hospital of Traditional Chinese Medicine (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Beijing Tiantan Hospital (Other); Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other); Hubei Zhongshan Hospital Affiliated to Wuhan University (Unknown)
Responsible Party: Sponsor-Investigator, Liu Hongfang, Chief Physician, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Other Study IDs: 2023ZD0509303-1
Record Dates: First submitted 2025-04-08; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Kidney Disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed group: People receiving exposure factors:In addition to the basic treatment and non-Yiqi Jiangzhuo Huoxue Tongluo Chinese patent medicine(except for Niaoduqing Granules, Shenshuaining Tablets/Capsules,Qizhi Capsules,Qizhi Yishen Capsules and other Chinese patent medicine),the exposure factors were treated with Shenqi Decoction(composed of Astragalus,Salvia miltiorrhiza,Leech,Rhubarb,Epimedium,Motherwort)as the representative of Yiqi Jiangzhuo Huoxue Tongluo Chinese medicine prescription treatment,and did not receive other traditional Chinese medicine treatment measures for urinary protein or renal insufficiency.The definition of basic treatment is:standardized diet,exercise,hypoglycemic,antihypertensive,lipid-lowering and other basic treatment measures,appropriate doses of angiotensin converting enzyme inhibitors(ACEI)/angiotensin receptor blockers(ARB),sodium-glucose co-transporter 2 inhibitors(SGLT2i),salt hormone receptor antagonists(MRA) and other drugs with clear renal protective effect
- Non-exposed group: Diabetic kidney disease patients who did not receive exposure factors.

SUMMARY:
In order to reduce the clinical demand for kidney dialysis rate of Diabetic Kidney Disease（DKD） patients, a bidirectional cohort study of 4472 patients with DKD (Qi deficiency and collateral stasis syndrome) was carried out based on a preliminary DKD cohort of 13,000 patients. The exposure factor was supplementing and reducing the kidney turbidity-Huoxue Tongluo method represented by the addition and subversion of Shenzhuo prescription, and the incidence of end-stage renal disease was the main therapeutic index. Follow-up was conducted for 2 years

ELIGIBILITY:
Inclusion Criteria:

* 1 in line with Western medicine diagnostic criteria for type 2 diabetic kidney disease ;
* 2 18-80 years old, regardless of gender ;
* 3 eGFR > 15ml / ( min · 1.73m2 ) ; the eGFR was calculated according to the chronic kidney disease epidemiology collaboration equation ( CKD-EPI ).
* 4 In line with the diagnostic criteria of qi deficiency and collateral stasis syndrome in traditional Chinese medicine ;
* 5glycosylated hemoglobin ( HbA1c ) between 7-10 % ;
* 6 blood pressure ≤ 160 / 100mmHg ;
* 7 to sign the informed consent ;

Exclusion Criteria:

* 1 combined with other clear renal diseases, such as polycystic kidney disease, glomerulonephritis, renal tumor, etc. ;
* 2 patients with a history of recurrent genitourinary tract infection ;
* 3 combined with cardiovascular and cerebrovascular, digestive, respiratory, urinary, immune system serious diseases or mental diseases ;
* 4 currently in pregnancy, lactation, or pregnancy plan women ;
* 5 Patients with type 1 diabetes.
* 6 Tumor patients undergoing radiotherapy, chemotherapy or targeted therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic kidney disease patients, in line with the inclusion criteria, do not meet the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 4472 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of end-stage renal disease | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  dialysis, transplantation or glomerular filtration rate ( eGFR ) < 15ml / ( min · 1.73m2 )

SECONDARY OUTCOMES:
Incidence of renal composite outcome indicators | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  End-stage renal disease [ dialysis, transplantation or glomerular filtration rate ( eGFR ) < 15ml / ( min · 1.73m2 ) ], eGFR decreased by more than 50 %, renal causes of death were defined.
Changes of urinary protein creatinine ratio | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Changes of urinary protein creatinine ratio
Changes of 24-hour urinary protein level | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Changes of 24-hour urinary protein level
Estimate the change value of glomerular filtration rate ( eGFR ) level, slope | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Estimate the change value of glomerular filtration rate ( eGFR ) level, slope
Chinese medicine syndrome scores | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  The TCM（Traditional Chinese Medicine） symptoms of the patients were scored by the TCM syndrome scale in order to judge the improvement of their symptoms.The highest score was 114 points, and the lowest score was 0 points. The higher the score, the worse the patient 's health.

OTHER OUTCOMES:
Body temperature | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Body temperature
blood pressure | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Both systolic and diastolic blood pressures should be measured.
respiration | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years.
  respiration
heart rate | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  heart rate
Number of participants with abnormal white blood cell count ( WBC ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal white blood cell count ( WBC )
Number of participants with abnormal electrocardiogram | Review period, enrollment, enrollment after two months, enrollment after half a year, enrollment after 1 year, enrollment after 1 and a half years, enrollment after two years
  Number of participants with abnormal electrocardiogram
glycosylated hemoglobin | Review period, enrollment, enrollment after two months, enrollment after half a year, enrollment after 1 year, enrollment after 1 and a half years, enrollment after two years
  glycosylated hemoglobin
fasting blood glucose | Review period, enrollment, enrollment after two months, enrollment after half a year, enrollment after 1 year, enrollment after 1 and a half years, enrollment after two years
  fasting blood glucose
incidence of adverse events | Review period, enrollment, enrollment after two months, enrollment after half a year, enrollment after 1 year, enrollment after 1 and a half years, enrollment after two years
  incidence of adverse events
Number of participants with abnormal red blood cell count ( RBC ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal red blood cell count ( RBC )
Number of participants with abnormal hemoglobin ( HGB ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal hemoglobin ( HGB )
Number of participants with abnormal lymphocyte percentage ( LY % ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal lymphocyte percentage ( LY % )
Number of participants with abnormal Percentage of neutrophils( NE % ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Percentage of neutrophils( NE % )
Number of participants with abnormal Platelet count ( PLT ) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Platelet count ( PLT )
Number of participants with abnormal Urine PH value | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urine PH value
Number of participants with abnormal Urinary protein | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urinary protein
Number of participants with abnormal Urine occult blood | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urine occult blood
Number of participants with abnormal Urinary glucose | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urinary glucose
Number of participants with abnormal Urine ketone | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urine ketone
Number of participants with abnormal Urine white blood cells (high magnification field of view) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urine white blood cells (high magnification field of view)
Number of participants with abnormal Urine red blood cells (high magnification field of view) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Urine red blood cells (high magnification field of view)
Number of participants with abnormal Serum alanine aminotransferase | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum alanine aminotransferase
Number of participants with abnormal Serum aspartate aminotransferase | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum aspartate aminotransferase
Number of participants with abnormal Serum alkaline phosphatase | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum alkaline phosphatase
Number of participants with abnormal Serum gamma-glutamyl transferase | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum gamma-glutamyl transferase
Number of participants with abnormal Serum albumin (ALB) | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum albumin (ALB)
Number of participants with abnormal Serum total bilirubin（TBIL） | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum total bilirubin（TBIL）
Number of participants with abnormal Serum direct bilirubin（DBIL） | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum direct bilirubin（DBIL）
Number of participants with abnormal Serum indirect bilirubin（IBIL） | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Number of participants with abnormal Serum indirect bilirubin（IBIL）
Serum urea | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Serum urea
Serum urate | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Serum urate
Serum cystatin C | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Serum cystatin C
Serum creatinine | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Serum creatinine
Plasma triglyceride | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Plasma triglyceride
Plasma high-density lipoprotein | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Plasma high-density lipoprotein
Plasma total cholesterol | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Plasma total cholesterol
Plasma low-density lipoprotein | Review period, enrollment, enrollment two months, enrollment half a year, enrollment 1 year, enrollment 1 and a half years, enrollment two years
  Plasma low-density lipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: HongFang Liu, Study Director — Dongzhimen Hospital
Locations (5):
- China (5):
  - Dongzhimen Hospital of BeijingUniversity of Chinese Medicine, Beijing, Beijing Municipality
  - Guang'anmen Hospital，China Academy of Chinese Medical Sciencescancel, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital to ChangChun University of Chinese Medicinecancel, Changchun, Jilin
  - Tianjin Medical University Chu Hsien-I Memorial Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No